CLINICAL TRIAL: NCT02702349
Title: The Frequency of Positive Challenge Test to Penicillin in Children Suspected to Have Allergy to Penicillin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 52-15
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): penicillin test and challenge
  Interventions: Other: penicillin test

INTERVENTIONS:
Other: penicillin test — children are tested for penicillin allergy and then challenged with penicillin P.O.

SUMMARY:
The incidence of reactions during penicillin challenge tests among children with suspected penicillin allergy

DETAILED DESCRIPTION:
children who are suspected to have penicillin allergy due to a suspected allergic reaction during penicillin treatment are sent for allergy investigation to role out allergy. Patients go through penicillin test and if negative are challenged by oral administration under medical observation. The investigators would like to check the incidence among our pediatric pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children older then 6 month with suspected penicillin allergy

Exclusion Criteria:

* Children under 6 month old

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of reactions during penicillin challenge tests among children with suspected penicillin allergy | one year
  To find out how many children are actually true allergic to penicillin

CONTACTS AND LOCATIONS:
Overall Officials: vered schichter- konfino, MD, Principal Investigator — Hillelyaffe medical center

IPD SHARING:
Plan to Share IPD: No